CLINICAL TRIAL: NCT02975661
Title: Registry of Huaier Granule for Prevention of Recurrence and Metastasis of Gastrointestinal Cancer After Radical Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Collaborators: Second Hospital of Jilin University (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: HE-201601
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Observational 1: Huaier Granule
- Observational 2: Radiotherapy or chemotherapy
- Observational 3: treatment abandoned
- Observational 4: Huaier Granule & Radiotherapy or chemotherapy

SUMMARY:
Registration of patients after gastrointestinal cancer radical surgery, including the information of treatments, recurrence & metastasis, adverse events,etc.

DETAILED DESCRIPTION:
This study adopts a multicenter, open, and registered research method, and plans to include 840 cases, including 360 cases in the Huaier Granule test group, 360 cases in the radiotherapy and chemotherapy control group, and 120 cases in the blank group. Using natural grouping, the registered objects are not pre grouped or queue divided, and the diagnosis, treatment, efficacy, and safety of gastrointestinal malignant tumor patients are accurately recorded under real conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gastrointestinal cancer (stomach, colon or rectum);
2. Patients who have received gastrointestinal cancer radical surgery within a month;
3. Patients between 18 and 70 years old,no gender restriction;
4. Patients volunteer to participate this study and have signed the informed consent form.

Exclusion Criteria:

1. No chemotherapy or combined radiation and chemotherapy indications；
2. Unable to cooperate to complete related information collection;
3. Participation in any other clinical trial within three months;
4. Conditions that are considered not suitable for this study investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after gastrointestinal cancer radical surgery.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 2 years
  Time from enrollment to tumor recurrence or death with any cause

SECONDARY OUTCOMES:
Disease situation | Baseline period
  Generally refers to tumor staging, classification, surgical methods, etc
Quality of Life Score | Up to 2 years
  Evaluate the quality of life of subjects during the trial by using the SF-36 scale.Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Postoperative treatment methods | Up to 2 years
  Generally including treatment plan, compliance, etc
Concomitant medication | Up to 2 years
  Other drugs (including chemical drugs, biological products, traditional Chinese patent medicines and simple preparations) taken by the subject in addition to the conventional research drugs during the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Tongjun Liu, PhD, Principal Investigator — Second Hospital of Jilin University
Locations (12):
- China (12):
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Qiqihar Medical College, Qiqihar, Heilongjiang
  - Hulunbuir People's Hospital, Hailar, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi